CLINICAL TRIAL: NCT06512961
Title: Applicability of Tissue Flossing for Blood Flow Restriction in the Upper Limb: Study of Reliability, Reproducibility and Performance Analysis
Brief Title: Applicability of Tissue Flossing for Blood Flow Restriction in the Upper Limb: Reliability and Performance Analysis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Principal Investigator, Franciele Marques Vanderle, Professor, Paulista University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 78229724.9.0000.5402
Record Dates: First submitted 2024-06-25; First posted 2024-07-22 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hypertrophy; Muscle Strength
Keywords: Tissue flossing; Blood flow restriction
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Traditional BFR (Active Comparator): This group will perform the training protocol with traditional BFR, using a pressure cuff as an occluder on both arms.
  Interventions: Device: Blood Flow Restriction Cuff; Other: Training Protocol
- Group BFR TF (Experimental): This group will perform the training protocol with BFR using TF on both arms.
  Interventions: Device: Tissue Flossing; Other: Training Protocol

INTERVENTIONS:
Device: Tissue Flossing — Tissue Flossing ia a elastic band that when applied exerts an external pressure above or below a muscle or joint of the extremities.
  Arms: Group BFR TF
Device: Blood Flow Restriction Cuff — Inflatable device that exerts an external pressure above a muscle or joint of the extremities.
  Arms: Group Traditional BFR
Other: Training Protocol — The upper limb resistance training protocol will follow that recommended in the study by Patterson et al. for resistance training, and will last 15weeks, with 3 training sessions per week, with a day break between sessions.

SUMMARY:
Blood flow restriction (BFR) is a widely studied technique that combines low-intensity exercise with vascular occlusion, resulting in muscular benefits. However, its application is challenging due to methodological variations and equipment costs. Tissue Flossing (TF) appears as an affordable alternative, but lacks solid scientific evidence.

DETAILED DESCRIPTION:
Objectives: to evaluate the intra- and inter-rater reliability of the occlusion pressure generated by TF, investigate the reproducibility of TF application on different days and compare TF with traditional RFS in terms of muscle gains.

Methods: the study is divided into two stages: First stage, randomized controlled crossover clinical trial, 80 healthy individuals aged 18 to 30 years old evaluated to determine the reliability of the TF. Participants will follow one of two types of randomization, with exclusions based on health criteria. Assessments include anthropometric characteristics, determination of occlusion pressure (POT), identification of 40% and 80% of POT, flow data and arterial diameter after TF application. Statistical analysis will use the intraclass correlation index (ICC) and specific models for intra- and inter-rater analyses. Second stage, randomized controlled clinical trial with parallel groups, 34 participants will be evaluated over fifteen weeks. The initial procedures involve anthropometric assessments, POT determination, myotonometry, ultrasound, perceptual scale and 1RM test, applied to both upper limbs. Participants will perform a upper limb training protocol using RFS or TF, following myotonometric and perceptual assessments. After training, final assessments will measure the same parameters initially assessed. Statistical analysis will use normality tests, Generalized Mixed Models and effect size analysis in SPSS software, with a significance level of p<0.05. Expected results: This study is expected to provide information on the reliability and reproducibility of TF in generating occlusion pressure. Furthermore, the investigatorsF seek to validate TF by comparing it with traditional RFS in terms of muscle gains. If effective, TF could become an affordable option to promote muscle gains, in different application scenarios.

Participants will be duly informed about the procedures and objectives of this study, and after agreeing, they will sign an informed consent form, effectively becoming part of it. In the consent form, participants will be asked if they agree to the use of their data if they choose to withdraw from the study. Participants will also be asked for permission for the research team to share relevant data with people at universities participating in the research or regulatory authorities, where relevant. The study were approved to the Research Ethics Committee of FCT/UNESP, Presidente Prudente, SP, Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who present one or more of the following characteristics will not be included:
* 1 presence of any health condition that contraindicates or prevents exercise;
* 2 diabetes and diagnosed high blood pressure;
* 3 inflammatory, psychiatric, cardiovascular and/or respiratory rheumatological disease; - -4 being dependent on alcohol, consuming drugs and/or being a smoker;
* 5 history of knee surgery (e.g., meniscal repair and ligament reconstruction) or recent upper limb musculoskeletal injury that may impair performance during tests or interventions (e.g., muscle injury, tendinopathy, patellofemoral pain and/or back pain column in the last six months);
* 6 use of ergogenic supplements to improve physical performance and/or muscle mass and/or vasoactive medications;
* 7 having one or more risk factors predisposing to thromboembolism

Exclusion Criteria:

* Participants will be excluded from the study if they:
* 1 have a health problem that does not allow them to continue;
* 2 wish to leave the study;
* 3 not sign the consent form

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Occlusion pressures (AOP, 80% and 40% of AOP) | 3 days
  To determine the AOP, the Doppler equipment transducer will be used, which will be positioned over the brachii artery to capture the auscultatory pulse. A blood pressure cuff will be fixed to the participant's thigh close to the region of the inguinal fold of the dominant limb, and then with the inflatable region of the cuff on the medial portion of the thigh covering the femoral artery, it will be progressively inflated, waiting 15 seconds every 30 mmHg until the point at which the auscultatory pulse of the brachii artery is interrupted.
Assessment of arterial flow and diameter | 3 days
  A Sonoline Sienna® vascular ultrasound will be used combined with a 40mm B-mode ultrasonic transducer with a 7.5 MHz linear beam, which will be coated with gel for acoustic contact and positioned longitudinally to the posterior brachii artery, enabling variables to be assessed. Doppler flow measurements of upper limb (peak systolic velocity [cm/s], end-diastolic velocity [cm/s] and arterial diameter).
Perceptual parameter | 3 days
  The perceptual parameter will be evaluated using a Borg CR10+ scale, representing the perception of discomfort, 0 represents no discomfort and 10 extremely uncomfortable.
Tissue Flossing Assessment | 3 days
  The application of tissue flossing on the leg will be carried out by always passing the elastic tape with 50% of the tape over the next strip, until the end of the elastic tape.
Weight | 3 days
  It will be collected with a weight balance
Height | 1 day
  It will be collected with a stadiometer
Body Fat | 1 day
  It will be collected with a adipometer
Arterial pressure | 1 day
  It will be collected with a sphygmomanometer
Perimetry of the dominant upper limb | 1 day
  It will be defined by the Waterloo Footedness
Limb length | 1 day
  Identified with a measuring tape
Perceived exertion scale | up to 15 weeks
  Adapted BORG scale, with 0 being "no effort" and 10 "maximum effort".
Method preference | up to 15 weeks
  Participants must answer a brief questionnaire about their preference for one of the BFR methods carried out, and justify why they chose it.
1 Maximum Repetition Test | up to 15 weeks
  The warm-up will include a series of 6 to 10 repetitions, using approximately 50% of the estimated load for the first attempt of the test (44). This warm-up will not only prepare participants but also familiarize them with the movement. The determination of the initial warm-up load will be made subjectively by the researcher responsible for the study, considering the participant's height, body mass and training experience as reference points (45).
  After the warm-up phase, up to five attempts will be given to find the 1RM, with intervals of 3 to 5 minutes between them (46). The load adjustment for subsequent attempts will be determined by the subjective perception of effort, according to the BORG scale, where the greater the perception of effort, the lower the percentage of load added for the next attempt. The 1RM will be established as the maximum load at which the participant can perform one repetition without compensation.
Myotonometry | up to 15 weeks
  Myotonometry will be assessed using the MyotonPRO® tool, which consists of a portable, wireless and non-invasive device.
  The measurement will be carried out once, and in each shot, the following myotonometry parameters will be calculated: the state of tension (tone) and biomechanical properties (rigidity and elasticity).
Ultrasound | up to 15 weeks
  The assessment of the muscular structure will be carried out using ultrasound images of the participant's upper limbs, which will be captured using BodyMetrix BX-2000.
  Participants will be assessed in the supine position with arms fully extended and muscles relaxed. The ultrasound transducer will be covered with water-soluble transmission gel and positioned perpendicular to the skin over the muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- UNESP, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No